CLINICAL TRIAL: NCT03902938
Title: Use of Biodesign® Otologic Graft in Canal Wall Down Mastoidectomy: A Prospective, Randomized Trial
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was stopped as the benefit was challenging to determine in the preliminary usage.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1322212
Record Dates: First submitted 2019-03-18; First posted 2019-04-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2022-08

CONDITIONS: Otologic Disease
MeSH Terms: conditions — Ear Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biodesign Otologic Graft (Experimental): Graft following canal wall down mastoidectomy.
  Interventions: Biological: Biodesign Otologic graft
- Autograft temporalis fascia (Active Comparator): Graft following canal wall down mastoidectomy.
  Interventions: Other: Autograft temporalis fascia

INTERVENTIONS:
Biological: Biodesign Otologic graft — Patient's mastoid cavity will be covered with porcine small intestine submucosa, Biodesign.
  Other Names: Porcine small intestine submucosa
  Arms: Biodesign Otologic Graft
Other: Autograft temporalis fascia — Patient's mastoid cavity will be covered with covered with autograft.
  Arms: Autograft temporalis fascia

SUMMARY:
This is a prospective, randomized trial to evaluate canal wall down mastoidectomy (CWDM) healing outcomes using Biodesign® small intestine submucosa graft compared to autologous temporalis fascia graft.

DETAILED DESCRIPTION:
Patients 18 or older will undergo primary canal wall down mastoidectomy. Patients with known biologic sensitivity or cultural objection to use of porcine materials will be excluded.

Data will be derived from the medical record and surgeon reports as detailed on pre-op and follow-up forms. Variables collected include age, gender, medical co-morbidities, body mass index, pre-operative audiometric values (including word recognition score, pure tone average, and air bone gap), side of surgery, size of operative cavity, infectious state (draining versus dry), exact surgical procedure, presence of cholesteatoma, time to dry cavity, time to complete epithelialization (as observed directly by the surgeon), and post-operative complications (such as persistent perforation, drainage, granulation tissue formation, and facial nerve outcomes). Dates and patient number will be recorded. Patients will be randomly assigned using randomization software, whereby patients will be assigned a sequential research number that is pre-randomized to one research arm. The study cannot be blinded, as the surgeon will be able to identify which graft will be used. De-identified photographs of the post-operative outcomes at each time point will be recorded photographically. Three physicians will review these photographs without prior knowledge of the treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary canal wall mastoidectomy

Exclusion Criteria:

* Patients with a known biologic sensitivity or a cultural aversion to the use of porcine materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Epithelialization of the canal wall down mastoid cavity | Evaluation at 1 month post-operatively.
  Direct observation by surgeon
Epithelialization of the canal wall down mastoid cavity | Evaluation at 2 months post-operatively.
  Direct observation by surgeon
Epithelialization of the canal wall down mastoid cavity | Evaluation at 3 months post-operatively.
  Direct observation by surgeon
Epithelialization of the canal wall down mastoid cavity | Evaluation at 6 months post-operatively.
  Direct observation by surgeon

SECONDARY OUTCOMES:
Determination of dry cavity | Evaluation at 1 month post-operatively
  Direct observation by surgeon
Determination of dry cavity | Evaluation at 2 months post-operatively
  Direct observation by surgeon
Determination of dry cavity | Evaluation at 3 months post-operatively
  Direct observation by surgeon
Determination of dry cavity | Evaluation at 6 months post-operatively
  Direct observation by surgeon
Audio-metric outcome | Evaluation at 3 months post-operatively
  Test the pure tone air conduction (average of 500, 1000 and 2000 Hz)
Audio-metric outcome | Evaluation at 3 months post-operatively
  Determine the Air Bone Gap by measuring the difference between the air conduction and bone conduction testing. The air bone gap is the difference between the 2 readings and must be present at 3 consecutive frequencies.
Audio-metric outcome | Evaluation at 3 months post-operatively
  The word recognition testing evaluates the patient's ability to repeat phonetically balanced words appropriate for their hearing level.
Audio-metric outcome | Evaluation at 6 months post-operatively
  Test the pure tone air conduction (average of 500, 1000 and 2000 Hz)
Audio-metric outcome | Evaluation at 6 months post-operatively
  Determine the Air Bone Gap by measuring the difference between the air conduction and bone conduction testing. The air bone gap is the difference between the 2 readings and must be present at 3 consecutive frequencies.
Audio-metric outcome | Evaluation at 6 months post-operatively
  The word recognition testing evaluates the patient's ability to repeat phonetically balanced words appropriate for their hearing level.

CONTACTS AND LOCATIONS:
Overall Officials: Seilesh Babu, MD, Principal Investigator — Physician of record
Locations (1):
- Ascension Providence Hospital, Novi Campus, Novi, Michigan, United States

REFERENCES:
- [Background] Ambro BT, Zimmerman J, Rosenthal M, Pribitkin EA. Nasal septal perforation repair with porcine small intestinal submucosa. Arch Facial Plast Surg. 2003 Nov-Dec;5(6):528-9. doi: 10.1001/archfaci.5.6.528. PMID 14623693
- [Background] Ansaloni L, Cambrini P, Catena F, Di Saverio S, Gagliardi S, Gazzotti F, Hodde JP, Metzger DW, D'Alessandro L, Pinna AD. Immune response to small intestinal submucosa (surgisis) implant in humans: preliminary observations. J Invest Surg. 2007 Jul-Aug;20(4):237-41. doi: 10.1080/08941930701481296. PMID 17710604
- [Background] Bejjani GK, Zabramski J; Durasis Study Group. Safety and efficacy of the porcine small intestinal submucosa dural substitute: results of a prospective multicenter study and literature review. J Neurosurg. 2007 Jun;106(6):1028-33. doi: 10.3171/jns.2007.106.6.1028. PMID 17564175
- [Background] Chhapola S, Matta I. Mastoid obliteration versus open cavity: a comparative study. Indian J Otolaryngol Head Neck Surg. 2014 Jan;66(Suppl 1):207-13. doi: 10.1007/s12070-011-0429-x. Epub 2012 Jan 1. PMID 24533385
- [Background] Gantz BJ, Wilkinson EP, Hansen MR. Canal wall reconstruction tympanomastoidectomy with mastoid obliteration. Laryngoscope. 2005 Oct;115(10):1734-40. doi: 10.1097/01.MLG.0000187572.99335.cc. PMID 16222186
- [Background] Illing E, Chaaban MR, Riley KO, Woodworth BA. Porcine small intestine submucosal graft for endoscopic skull base reconstruction. Int Forum Allergy Rhinol. 2013 Nov;3(11):928-32. doi: 10.1002/alr.21206. Epub 2013 Aug 16. PMID 23956139
- [Background] Kanazawa Y, Shojaku H, Okabe M, Fujisaka M, Takakura H, Tachino H, Tsubota M, Watanabe Y, Nikaido T. Application of hyperdry amniotic membrane patches without fibrin glue over the bony surface of mastoid cavities in canal wall down tympanoplasty. Acta Otolaryngol. 2012 Dec;132(12):1282-7. doi: 10.3109/00016489.2012.701329. Epub 2012 Nov 6. PMID 23126613
- [Background] Knoll LD. Use of porcine small intestinal submucosal graft in the surgical management of Peyronie's disease. Urology. 2001 Apr;57(4):753-7. doi: 10.1016/s0090-4295(00)01079-7. PMID 11306396
- [Background] Kobayashi T, Gyo K, Komori M, Hyodo M. Polyglycolic acid sheet attached with fibrin glue can facilitate faster epithelialization of the mastoid cavity after canal wall-down tympanoplasty. Auris Nasus Larynx. 2017 Dec;44(6):685-689. doi: 10.1016/j.anl.2017.01.013. Epub 2017 Feb 20. PMID 28215637
- [Background] Lin HK, Godiwalla SY, Palmer B, Frimberger D, Yang Q, Madihally SV, Fung KM, Kropp BP. Understanding roles of porcine small intestinal submucosa in urinary bladder regeneration: identification of variable regenerative characteristics of small intestinal submucosa. Tissue Eng Part B Rev. 2014 Feb;20(1):73-83. doi: 10.1089/ten.TEB.2013.0126. Epub 2013 Jul 25. PMID 23777420
- [Background] Martini A, Morra B, Aimoni C, Radice M. Use of a hyaluronan-based biomembrane in the treatment of chronic cholesteatomatous otitis media. Am J Otol. 2000 Jul;21(4):468-73. PMID 10912689
- [Background] Murphy F, Corbally MT. The novel use of small intestinal submucosal matrix for chest wall reconstruction following Ewing's tumour resection. Pediatr Surg Int. 2007 Apr;23(4):353-6. doi: 10.1007/s00383-007-1882-1. Epub 2007 Feb 8. PMID 17287942
- [Background] Ort SA, Ehrlich HP, Isaacson JE. Acellular porcine intestinal submucosa as fascial graft in an animal model: applications for revision tympanoplasty. Otolaryngol Head Neck Surg. 2010 Sep;143(3):435-40. doi: 10.1016/j.otohns.2010.04.268. PMID 20723784
- [Background] Palva T. Surgical treatment of chronic middle ear disease. II. Canal wall up and canal wall down procedures. Acta Otolaryngol. 1987 Nov-Dec;104(5-6):487-94. doi: 10.3109/00016488709128279. PMID 3434271
- [Background] Rutner AB, Levine SR, Schmaelzle JF. Processed porcine small intestine submucosa as a graft material for pubovaginal slings: durability and results. Urology. 2003 Nov;62(5):805-9. doi: 10.1016/s0090-4295(03)00664-2. PMID 14624898
- [Background] Seymour PE, Leventhal DD, Pribitkin EA. Lip augmentation with porcine small intestinal submucosa. Arch Facial Plast Surg. 2008 Jan-Feb;10(1):30-3. doi: 10.1001/archfacial.2007.17. PMID 18209120
- [Background] Sheehy JL. Cholesteatoma surgery: canal wall down procedures. Ann Otol Rhinol Laryngol. 1988 Jan-Feb;97(1):30-5. doi: 10.1177/000348948809700106. PMID 3277524
- [Background] Spiegel JH, Kessler JL. Tympanic membrane perforation repair with acellular porcine submucosa. Otol Neurotol. 2005 Jul;26(4):563-6. doi: 10.1097/01.mao.0000169636.63440.4e. PMID 16015147
- [Background] Wetmore SJ, Bueller HA, Cost JL. Split thickness skin grafting in canal wall down tympanomastoidectomy. Otol Neurotol. 2014 Jan;35(1):97-100. doi: 10.1097/MAO.0b013e3182a4445d. PMID 24136321